CLINICAL TRIAL: NCT01790152
Title: Health Effects After Anthracycline and Radiation Therapy (HEART): Dexrazoxane and Prevention of Anthracycline-Related Cardiomyopathy
Brief Title: Effects of Dexrazoxane Hydrochloride on Biomarkers Associated With Cardiomyopathy and Heart Failure After Cancer Treatment
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE11C2; S0004187 (CTRP (Clinical Trial Reporting Program)); ALTE11C2 (Other: Childrens Oncology Group); COG-ALTE11C2 (Other: DCP); ALTE11C2 (Other: CTEP); R01CA211996 (NIH); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hodgkin Lymphoma in Remission; Leukemia in Remission; Lymphoblastic Lymphoma; Osteosarcoma; Recurrent Leukemia; Recurrent Lymphoma; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteosarcoma; Leukemia; Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (laboratory biomarker analysis): Patients complete a diagnostic symptom checklist, undergo a physical exam, echocardiogram, collection of serum for biomarker testing, and a 6 minute walk test, and complete quality of life, family history, physical activity, and smoking questionnaires.
  Interventions: Other: Assessment of Therapy Complications; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Assessment of Therapy Complications — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effects of dexrazoxane hydrochloride on biomarkers associated with cardiomyopathy and heart failure after cancer treatment. Studying samples of blood in the laboratory from patients receiving dexrazoxane hydrochloride may help doctors learn more about the effects of dexrazoxane hydrochloride on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether leukemia and lymphoma patients from P9404, P9425, P9426, and Dana Farber Cancer Institute (DFCI) 95-01 randomized to the experimental dexrazoxane hydrochloride (DRZ) arms have decreased markers of cardiomyopathy/heart failure (CHF) compared with patients on the standard arm.

II. To determine whether osteosarcoma patients from P9754 (all received DRZ) have decreased markers of cardiomyopathy/heart failure (CHF) compared with similarly treated osteosarcoma patients diagnosed during the same time period, but who did not receive DRZ.

III. To evaluate whether the cardioprotective effect of DRZ is modified by anthracycline (anthracycline analogue GPX-150) dose, chest radiation, and demographic factors (age at cancer diagnosis, current age, sex).

SECONDARY OBJECTIVES:

I. To determine whether leukemia and lymphoma patients from P9404, P9425, P9426, and DFCI 95-01 on the DRZ arms experienced differential rates of overall-survival and event-free survival compared with the standard therapy arms.

II. To determine whether projected quality-adjusted life years (QALY) differed by DRZ status, accounting for premature cardiac disease, primary disease relapse, and second cancers.

III. Determine the longitudinal trajectory of 2-dimensional echocardiographic parameters (focusing on left ventricular [LV] function and remodeling/geometric changes that can be reliably re-measured) among patients from time of cancer treatment through subsequent follow-up.

OUTLINE:

Patients complete a diagnostic symptom checklist, undergo a physical exam, echocardiogram, collection of serum for biomarker testing, and a 6 minute walk test, and complete quality of life, family history, physical activity, and smoking questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Study Strata I, II, and III are closed for further patient entry as of March 31, 2021. The study remains open for existing medical record submission of Stratum IV

* STRATUM I AND STRATUM II: LEUKEMIA AND LYMPHOMA SURVIVORS
* Previously enrolled leukemia and lymphoma survivors, randomized to + or - DRZ on P9404, P9425, P9426, or DFCI 95-01 (high-risk patients only)
* STRATUM I: Alive and in continuous first complete remission from their original cancer (leukemia/lymphoblastic lymphoma [P9404, high-risk DFCI 95-01] or Hodgkin lymphoma [P9425/P9426])
* STRATUM I: Did not have progressive disease or induction failure requiring off-protocol therapy including hematopoietic cell transplantation
* STRATUM I: Must not have been diagnosed with any subsequent malignancy that required additional cardiotoxic therapies (i.e., radiotherapy to the chest [also includes fields directed towards the neck, upper abdomen, or spine], or additional anthracyclines or anthraquinones); patients with history of subsequent malignancy that did not require such therapies remain eligible
* STRATUM I: All patients and/or their parents or legal guardians must sign a written informed consent
* STRATUM II: Among leukemia and lymphoma patients randomized to + or - DRZ on P9404, P9425, P9426, and DFCI 95-01 (high risk patients only) who have relapsed or have experienced a subsequent malignancy that precludes eligibility since their original diagnosis, the study committee will review the available data (both from Children's Oncology Group's [COG?s] Statistics and Data Center [SDC] and the participating institution) to determine if individual patients are to be selected for Stratum 2; in recognition that local institutions sometimes have more updated relapse/subsequent cancer data than SDC, in cases where local data is more updated, local data will be used preferentially; the study will petition the Institutional Review Board (IRB) specifically for a waiver of consent to include any relapse and subsequent cancer data obtained from existing records for analysis of the secondary aims; patients selected for Stratum 2 will be those for whom late relapse or subsequent cancer is reported but who lack clear confirmation in existing records (either at SDC or at the local institution)
* STRATUM II: Alive, but have experienced relapse of their original cancer and/or have developed a subsequent cancer (other than non-melanomatous skin cancer) since their original diagnosis
* STRATUM II: All patients and/or their parents or legal guardians must sign a written informed consent
* STRATUM III: OSTEOSARCOMA SURVIVORS
* Previously enrolled osteosarcoma survivors treated on P9754 who are alive and able (themselves and/or parents/legal guardian) to provide written informed consent; note that relapse and subsequent malignancy are not exclusion criteria for P9754 survivors
* Comparison subjects for P9754 survivors will be eligible to be enrolled from any ALTE11C2 participating COG site (even if that institution did not participate on P9754), according to the following criteria:

  * Newly diagnosed, previously untreated biopsy-proven moderate or high grade osteosarcoma without metastasis; patients with low grade osteosarcoma, parosteal or periosteal sarcoma are ineligible
  * < 31 years of age at time of initial osteosarcoma diagnosis
  * Diagnosis occurred between January 1, 1999 through December 31, 2002; duration of therapy can extend beyond 2002
  * No evidence of poor or low cardiac function at time of initial osteosarcoma diagnosis; if reports from the time are available: shortening fraction >= 28% by echocardiogram and within the institutional normative range for age, or radionuclide angiogram ejection fraction >= 50%; if imaging reports from the time are no longer available, there must be no documentation within available medical records that suggest poor or low cardiac function at time of diagnosis
  * Comparison subject must have institutional records (e.g., clinic note, treatment summary, chemotherapy roadmap) documenting lifetime receipt of 450 to 600 mg/m^2 of doxorubicin (doses within 10% are acceptable); this includes initial therapy as well as any subsequent therapy for relapse or second cancer, if relevant; as such, comparison subjects who have had osteosarcoma relapse or subsequent malignancies remain eligible so long as they meet all other eligibility criteria
  * No anthracycline or anthraquinone aside from doxorubicin was ever given as part of initial or subsequent therapies
  * No exposure to DRZ at any point in time
  * All patients and/or their parents or legal guardians must sign a written informed consent
* STRATUM IV: CARDIOMYOPATHY CASES, NOT OTHERWISE ELIGIBLE FOR STRATUMS 1, 2, AND 3
* Individuals diagnosed with cancer prior to age 21 years, who required treatment with chemotherapy and/or radiotherapy, achieved initial remission, and remained alive after completing anti-cancer-therapy for at least 1 year
* Must have screening echocardiograms for heart function as part of cancer therapy and off-therapy evaluations available (Digital Imaging and Communications in Medicine [DICOM] format). Images from Video Home System (VHS) tapes and reports only (without images) are not suitable
* Cannot have a known history of congenital heart disease (patent foramen ovale remain eligible) or underlying genetic syndrome associated with abnormal cardiovascular development or health (e.g., down syndrome)
* Based on echocardiography, must have either left ventricular fractional shortening =< 28.0% or ejection fraction =< 50.0% on at least two occasions, with at least one of these measurements occurring after cancer therapy completion and be in the absence of sepsis or any uncontrolled infection
* If the fractional shortening or ejection fraction criteria is only met on one occasion, this must be after cancer therapy completion, be in the absence of sepsis or any uncontrolled infection, and the patient must have subsequently started on chronic medical therapy for cardiomyopathy (e.g., beta-blocker, angiotensin-converting enzyme [ACE]-inhibitor, angiotensin receptor blocker) lasting at least 6 months
* For all participants (stratums 1, 2, 3, and 4), all institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with leukemia or lymphoma enrolled on Pediatric Oncology Group (POG) P9404, P9425, P9426, and DFCI 95-01 or osteosarcoma enrolled on P9754
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2014-03-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular function and measures of pathologic remodeling (i.e., thickness-to-dimension ratio) assessed using standard 2-dimensional, M-mode, and Doppler echocardiogram | Baseline
  Univariate tests will be used as well as examination of the entire cohort via multivariable regression adjusting for all a priori covariates of interest.
Differences in serum biomarkers (particularly cardiac troponins and natriuretic peptides) | Baseline
  Univariate tests will be used as well as examination of the entire cohort via multivariable regression adjusting for all a priori covariates of interest.

SECONDARY OUTCOMES:
Quality of life based on self-report instruments | Baseline
  An analytic Markov model will be created and used. Estimates and their 95% confidence will be included to explore the sensitivity of any quality-adjusted life years estimates.
Primary disease relapse | Baseline
  An analytic Markov model will be created and used.
Second cancer rates | Baseline
  An analytic Markov model will be created and used.
Longitudinal trajectory of 2-dimensional echocardiographic parameters | From time of cancer treatment to subsequent follow-up
  Will utilize generalized linear model-general estimation equation to model the trajectories of echocardiographic biomarker estimates (continuous outcomes) across time. Relevant model shapes will be evaluated, beginning with linear models, but also testing more flexible shapes (e.g., quadratic, cubic, or cubic spline functions with varying numbers of knots) to determine whether non-linear components are needed for fit. Will also examine interactions of dexrazoxane (DRZ) status with the selected functions of time to evaluate for differences in trajectories over time by DRZ status.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Chow, Principal Investigator — Children's Oncology Group
Locations (79):
- United States (69):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Chow EJ, Aggarwal S, Doody DR, Aplenc R, Armenian SH, Baker KS, Bhatia S, Blythe N, Colan SD, Constine LS, Freyer DR, Kopp LM, Laverdiere C, Leisenring WM, Sasaki N, Vrooman LM, Asselin BL, Schwartz CL, Lipshultz SE. Dexrazoxane and Long-Term Heart Function in Survivors of Childhood Cancer. J Clin Oncol. 2023 Apr 20;41(12):2248-2257. doi: 10.1200/JCO.22.02423. Epub 2023 Jan 20. PMID 36669148
- [Result] Lipshultz ER, Chow EJ, Doody DR, Armenian SH, Asselin BL, Baker KS, Bhatia S, Constine LS, Freyer DR, Kopp LM, Schwartz CL, Lipshultz SE, Vrooman LM. Cardiometabolic Risk in Childhood Cancer Survivors: A Report from the Children's Oncology Group. Cancer Epidemiol Biomarkers Prev. 2022 Mar 1;31(3):536-542. doi: 10.1158/1055-9965.EPI-21-0360. PMID 34810210
- [Result] Chow EJ, Aplenc R, Vrooman LM, Doody DR, Huang YV, Aggarwal S, Armenian SH, Baker KS, Bhatia S, Constine LS, Freyer DR, Kopp LM, Leisenring WM, Asselin BL, Schwartz CL, Lipshultz SE. Late health outcomes after dexrazoxane treatment: A report from the Children's Oncology Group. Cancer. 2022 Feb 15;128(4):788-796. doi: 10.1002/cncr.33974. Epub 2021 Oct 13. PMID 34644414
- [Derived] Chow EJ, Asselin BL, Schwartz CL, Doody DR, Leisenring WM, Aggarwal S, Baker KS, Bhatia S, Constine LS, Freyer DR, Lipshultz SE, Armenian SH. Late Mortality After Dexrazoxane Treatment: A Report From the Children's Oncology Group. J Clin Oncol. 2015 Aug 20;33(24):2639-45. doi: 10.1200/JCO.2014.59.4473. Epub 2015 May 26. PMID 26014292